CLINICAL TRIAL: NCT00427362
Title: A Canadian Open-Label Study to Evaluate the Safety and Effectiveness of Adalimumab When Added to Inadequate Therapy for the Treatment of Psoriatic Arthritis (PsA) (ACCLAIM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W05-399; ACCLAIM
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2008-04

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
To further assess the safety and effectiveness of adalimumab 40mg in the treatment PsA who have had an unsatisfactory response or intolerance to prior or ongoing DMARDs

ELIGIBILITY:
Inclusion Criteria:

* Active psoriatic arthritis defined by >= 3 tender or painful joints and >= 3 swollen joints despite standard psoriatic arthritis therapy
* Has had an unsatisfactory response or intolerance to at least two prior or ongoing DMARDs (one of which has to be methotrexate)

Exclusion Criteria:

* Has a history of cancer or other than certain skin or cervical cancers
* Has a history of, or current acute inflammatory joint disease of origin other than PsA, e.g., systemic lupus erythematosus etc.
* Has other, unstable diseases, including congestive heart failure, inflammatory bowel disease, recent stroke, leg ulcers or other condition which would put the subject at risk
* History of active tuberculosis, history of histoplasmosis or listeriosis
* Latent TB or risk factors for the activation of latent TB, e.g. previous exposure to TB, and has not initiated TB prophylaxis prior to the first adalimumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
ACR20 response | Week 12

SECONDARY OUTCOMES:
ACR50 | Week 12
ACR70 | Week 12
PsARC | Week 12
DAS28 | Week 12
PASI50/75 | Week 12
HAQ-DI | Week 12
PsAQoL | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Guerette, PhD, Study Director — Abbott

REFERENCES:
- [Derived] Gladman DD; ACCLAIM Study Investigators; Sampalis JS, Illouz O, Guerette B. Responses to adalimumab in patients with active psoriatic arthritis who have not adequately responded to prior therapy: effectiveness and safety results from an open-label study. J Rheumatol. 2010 Sep;37(9):1898-906. doi: 10.3899/jrheum.100069. Epub 2010 Jul 1. PMID 20595284